CLINICAL TRIAL: NCT03209232
Title: Infliximab Accelerated Induction for Moderate to Severe Ulcerative Colitis in Children (INDUCE) Trial
Brief Title: Infliximab Accelerated Induction in Moderate to Severe Pediatric UC
Acronym: INDUCE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty to recruit patients and as high dose infliximab for severe UC is now the rule rather than the exception
Sponsor: Schneider Children's Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Amit Assa, Head of IBD program, Schneider Children's Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INDUCE
Record Dates: First submitted 2017-07-01; First posted 2017-07-06 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Accelerated induction (Experimental): Patients in group 1 will receive an accelerated induction of infliximab at 0,1,3 weeks (5 mg/kg) and then at week 7,11,15.
  Interventions: Drug: Infliximab
- Per protocol (Active Comparator): Patients in group 2 will receive a per protocol induction of infliximab at 0,2,6 weeks (5 mg/kg) and then at week 14.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Accelerated induction of infliximab in moderate to severe ambulatory prdiatric UC patients

SUMMARY:
Objectives: To examine the effect of accelerated infliximab induction in children with moderate to severe UC. Design: A multi-center, prospective, randomized, open label study. Setting: Pediatric gastroenterology centers. Participants: Children 6 year to 17 years (Overall, 84 patients) with moderate to severe UC who are corticosteroid dependent/resistant thus planned to receive infliximab induction. Intervention: Group 1 (intervention) will receive an accelerated induction at 0,1,3 weeks (5 mg/kg) and then at week 7,11,15. Group 2 (standard) will receive a per protocol induction at 0,2,6 weeks (5 mg/kg) and then at week 14. Drug levels will be obtained prior to each infusion in each group (up to week 20). Further maintenance will be planned according to drug levels at weeks 15 and 14, respectively. Follow-up will continue without further interventions till 52 weeks following induction. Main outcome measure: Clinical remission, on infliximab at week 20. Secondary outcome measures: 1. Colectomy free rates at week 20 and 52. 2. Clinical remission on infliximab at week 52. 3. Drug levels and anti-drug antibodies prior to last study infusion. 4. Anthropometric and laboratory measures including calprotectin at the end of induction, week 20 and week 52 5. Changes in fecal microbiome, virome and bile acids content. Sample size: In order to demonstrate 30% difference in clinical remission rate between groups is significant, we will need to study 36 children in each group to be able to reject the null hypothesis that the failure rates between the groups are equal with probability (power) of 80% and a type I error probability of 0.05.

DETAILED DESCRIPTION:
General intervention scheme:

The decision to start IFX is the sole decision of the treating physician based on the patient's immediate need. Eligible patients are those who are planned to start IFX. All patients will undergo clinical and laboratory evaluation for IFX eligibility (PPD, infectious serology). If the tests have already done in the last 3 months, we will use these data, there is no need to repeat. Patients must have a negative stool culture, stool for parasites and clostridium difficile toxin test performed over the last week in order to be eligible. The screening visit may be performed concomitantly with the enrolment visit if all inclusion and exclusion criteria are met.

Patients will be enrolled at the first screening visit. Informed consent will be signed by both parents is required during enrollment. Informed assent will be offered for patients 14 years old and older. Eligible patients, ambulatory UC patients, requiring IFX for corticosteroid dependent or refractory moderate to severe disease (excluding acute severe UC), meeting inclusion/exclusion criteria, after obtaining informed consent, will be randomized (1:1 ratio in blocks of four, stratified by immunomodulators use) at enrollment visit (week 0, prior to IFX initiation) to either group 1 or group 2 using opaque, numbered and sealed envelopes. Prior corticosteroid treatment is allowed as a taper-down schedule during induction with IFX and must be terminated by week 10 (otherwise will be defined as induction failure). At each visit all patients will be examined and have height, weight, and PUCAI performed as well as comprehensive laboratory examinations including CBC, albumin, AST, ALT, ESR and CRP (CRP will be measured and registered in mg/dL) and fecal samples (4 grams) for bile acids and microbiome/virome. Fecal sample for fecal calprotectin (FC) will be obtained as well at weeks 20 and 52. Extent of disease will be registered using the Paris classification (Levine A et al, IBD, June 2011) and will be based on the latest colonoscopic evaluation (described only by macroscopic involvement). Patients who undergo a colonoscopy at any time as standard of care before initiating biologic therapy should register the results of colonoscopy (according to the Mayo score- A score of ≤1 is considered complete mucosal healing). In addition, every colonoscopy that will be performed during the study period based on physician discretion, should be register in the CRF (Colonoscopy is not part of this specific protocol).

The study period is composed of two distinctive phases: Intervention phase: week 0-20 and follow-up phase: week 21-52.

Group 1 (intervention group): Patients in group 1 will receive an accelerated induction at 0,1,3 weeks (5 mg/kg) and then at week 7,11,15.

Group 2 (control group): Patients in group 2 will receive a per protocol induction at 0,2,6 weeks (5 mg/kg) and then at week 14.

Intensification by shortening intervals between infusion rather than dose increment was chosen based on the pharmacokinetics of IFX in severe disease favoring this strategy in-order to maintain adequate trough drug-levels and avoid intermittent exposure (23).

Drug levels will be obtained prior to each infusion in each group in the intervention phase. Further maintenance will be planned according to drug levels at weeks 15 and 14, respectively. A visit concluding the intervention phase will be performed at week 20. The follow-up phase will continue without further interventions till week 52. During the follow-up phase (maintenance) treatment will be administered according to the treating physician discretion, with no restrictions.

Patients with induction failure in the control arm (defined as a lack of improvement of at least 20 points from the baseline PUCAI score OR PUCAI≥35 at 3 weeks following induction) will be able to undergo treatment intensification by decreasing infusion intervals according to the treating physician discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Ulcerative colitis
2. PUCAI≥35
3. Age: 6 - 17 years (inclusive)
4. Planned to initiate IFX therapy.
5. Naïve to biologics
6. Informed consent
7. Neg. PPD-Test, negative HBV- S Ag
8. Negative stool culture, parasites and clostridium toxin

Exclusion Criteria:

1. Pregnancy.
2. Acute severe colitis.
3. Renal Failure.
4. Toxic megacolon.
5. Patients whose disease is confined to the rectum (i.e. proctitis).
6. Prior treatment with infliximab or adalimumab.
7. Previous malignancy.
8. Sepsis or active bacterial infection.
9. Known immune deficiency.
10. Positive Hepatitis B surface antigen or evidence for TB.
11. IBD unclassified.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Clinical remission on infliximab | 20 weeks
  The proportion of patients treated with infliximab in complete clinical remission (PUCAI<10)

SECONDARY OUTCOMES:
Colectomy free rate | 52 weeks
  The proportion of patients who did not underwent surgery
Clinical remission on infliximab | 52 weeks
  The proportion of patients treated with infliximab in complete clinical remission (PUCAI<10)
Drug levels prior to last study infusion | 14 weeks
  Infliximab level (microgram per mililiter) at the end of induction
Calprotectin level | 20 weeks
  Level of fecal calprotectin (microgram per gram)
Adverse events | 20 weeks
  The rate of drug related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Amit Assa, MD, Principal Investigator — Schneider Children's Medical Center, Israel
Locations (1):
- Schenider Children's Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No